CLINICAL TRIAL: NCT01493869
Title: A Phase I, Open-Label, Parallel-Group, Single-Dose Study to Assess the Pharmacokinetics of XL184 (Cabozantinib) Capsules in Hepatic Impaired Adult Subjects
Brief Title: Study to Assess the Pharmacokinetics of Cabozantinib (XL184) in Hepatic Impaired Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XL184-003
Record Dates: First submitted 2011-10-11; First posted 2011-12-16 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2014-09

CONDITIONS: Healthy; Hepatic Impairment
Keywords: Normal healthy adult subjects; Adult subjects with hepatic impairment
MeSH Terms: interventions — cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (Experimental): Subjects with normal hepatic function: healthy normal adult subjects
  Interventions: Drug: cabozantinib
- Group 2 (Experimental): Subjects with mild hepatic impairment: adult subjects with a Child-Pugh grade A (score 5-6).
  Interventions: Drug: cabozantinib
- Group 3 (Experimental): Moderate hepatic impairment: adult subjects with a Child-Pugh grade B (score 7-9).
  Interventions: Drug: cabozantinib
- Group 4 (Experimental): Severe hepatic impairment: adult subjects with a Child-Pugh grade C (score 10-15).
  Interventions: Drug: cabozantinib

INTERVENTIONS:
Drug: cabozantinib — 3 25-mg strength capsules (75-mg dose) administered as a single oral dose on Day 1 of study participation
  Other Names: XL184

SUMMARY:
The main objective of this study is to compare the pharmacokinetics (PK) of a single oral 75 mg dose of cabozantinib in hepatic impaired adult subjects to healthy adult subjects. Another objective is to assess the safety and tolerability of cabozantinib in these adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body weight must be ≥50 kg and <130 kg with a BMI of ≥18 (kg/m2) and ≤36.0 (kg/m2).
* Must use acceptable forms of birth control during the course of the study and for 3 months following the single dose of study drug.
* Female subjects of childbearing potential must have a negative pregnancy test at screening and check-in.
* Must have adequate vital sign reads at screening and check-in.
* Must be able to comply with dietary and fluid restrictions required for the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-09; Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
AUC, Cmax, tmax, t1/2, CL/F, and V/F parameters as a measure of the PK of a single oral 75 mg dose of cabozantinib in hepatic impaired adult subjects compared to healthy adult subjects matched for age, gender, body mass index (BMI), and ethnicity | Days 1 - 5, 6, 8, 11, 15, 19, 21, and 22
  Subjects will receive a single oral 75 mg dose of cabozantinib on Day 1 and then undergo periodic assessments Days 1 through 5 following this single dose, as well as on the mornings of Days 6, 8, 11, 15, 19, 21, and 22.

SECONDARY OUTCOMES:
Number of participants with adverse events, serious adverse events, and laboratory abnormalities as a measure of the safety and tolerability of a single oral 75 mg dose in hepatic impaired adult subjects and healthy adult subjects | Days 1 - 5, 6, 8, 11, 15, 19, 21, and 22

CONTACTS AND LOCATIONS:
Locations (1):
- McGuire VA Medical Center, Richmond, Virginia, United States